CLINICAL TRIAL: NCT06555133
Title: A Phase II Pilot Study of yttriuM-90 in Combination With capEcitabine and aTezolizumab for oligomEtastatic cOlorectal Cancer With unResectable lIver MeTastasEs (METEORITE)
Brief Title: Y-90, Capecitabine, and Atezolizumab for Oligometastatic CRC
Acronym: METEORITE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Sirtex Medical (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 430
Record Dates: First submitted 2024-05-02; First posted 2024-08-15 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Carcinoma Metastatic in the Liver
MeSH Terms: interventions — Capecitabine; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- yttriuM-90 in combination with capEcitabine and aTezolizumab (Experimental): Atezolizumab 1,200 mg IV every 3 weeks for 5 doses Capecitabine 825 mg/m2 PO BID for 2 weeks beginning on the date of each Y-90 therapy administration Y-90 radioembolization one or both hemilivers based on distribution of disease
  Interventions: Combination Product: yttrium-90 radioembolization

INTERVENTIONS:
Combination Product: yttrium-90 radioembolization — yttrium-90 radioembolization in combination with capecitabine and atezolizumab for the treatment of unresectable colorectal cancer liver metastases in individuals who have been treated with two or more lines of systemic therapy.
  Other Names: capecitabine and atezolizumab

SUMMARY:
BrUOG-430 is a prospective, single-arm, phase 2 trial evaluating yttrium-90 radioembolization in combination with capecitabine and atezolizumab for the treatment of unresectable colorectal cancer liver metastases in individuals who have been treated with two or more lines of systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of colorectal adenocarcinoma
2. Surgically unresectable, liver-isolated or liver-dominant, RECIST measurable, metastatic disease
3. Age ≥18 years at the time of signing informed consent
4. ECOG performance status 0 or 1
5. Progression on 2 or more lines of systemic therapy
6. Agreeable to providing tumor tissue and blood for exploratory correlative analyses
7. Less than 50% of liver volume replaced by metastatic disease (as determined by investigator)
8. Demonstrate adequate organ function as defined in table below (all screening labs should be performed within 14 days of atezolizumab initiation):

   Hematologic Absolute neutrophil count (ANC) ≥1,500 /mcL or ≥1,200 /mcL for those with benign ethnic neutropenia Absolute Lymphocyte Count (ALC) ≥ 0.5 x 109/L (500/uL) Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L within 7 days of assessment. Patient may be transfused or receive EPO to meet this criterion

   Renal Serum creatinine OR measured or calculated creatinine clearance ≤1.5 X upper limit of normal (ULN) OR (GFR can also be used in place of creatinine or CrCl) ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN

   Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 5 X ULN Alkaline Phosphatase ≤ 5 X ULN Albumin ≥2.5 mg/dL

   Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen

   ≤1.5 X ULN unless subject is receiving anticoagulant therapy. For patients receiving therapeutic anticoagulation: stable anticoagulant regimen

   Creatinine clearance should be calculated per institutional standard. Exceptions can be made for patients with known Gilbert disease (≤ 3X ULN)
9. Female subjects of childbearing potential must be willing to use an adequate method of contraception from the time of the negative pregnancy test until a minimum of 6 months after the last dose of study drug. Effective forms of contraception include abstinence, hormonal contraceptive (injectable or implantable), or intrauterine device in conjunction with a barrier method. Breast feeding subjects must be willing to discontinue at treatment start and for 5 months post-treatment.
10. Male subjects of childbearing potential must agree to use an adequate method of contraception with female partners of childbearing potential including abstinence or condoms plus an additional contraceptive method such as hormonal contraceptive (injectable or implantable), or intrauterine device during the study and for up to 3 months after the last dose of study drug.
11. Ability to understand and the willingness to sign a written informed consent document and to comply with the study protocol procedures

Exclusion Criteria:

1. Prior yttrium-90 therapy
2. Prior external beam radiation therapy to the liver
3. Predicted life expectancy of less than 3 months
4. Known mismatch repair deficiency (dMMR), microsatellite instability (MSI-H), or high tumor mutational burden (TMB-H) defined as ≥ 10 mutations per megabase
5. Known metastasis to the peritoneum or central nervous system. Exceptions include subjects with untreated brain metastases ≤ 1 cm, if asymptomatic and not requiring immediate radiation or steroids, and subjects with brain metastases that are treated and stable for 1 month
6. Treatment with investigational therapy within the 28 days of initiation of study treatment
7. Systemic treatment within 14 days or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
8. Prior treatment with CD137 agonists or anti-PD1, anti-PD-L1, anti-CTLA4 antibodies
9. A history of or current evidence of any condition (e.g. known deficiency of the enzyme dihydropyrimidine dehydrogenase [DPD]), therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
10. Known New York Heart Association class 3/4 congestive heart failure, left ventricular ejection fraction <40% (if previously measured), myocardial infarction within 6 months prior to enrollment, unstable angina, or unstable arrhythmia
11. Chronic obstructive pulmonary disease (COPD) requiring oral corticosteroids or chronic oxygen
12. History of autoimmune disease, including, but not limited to myasthenia gravis, myositis, autoimmune hepatitis, idiopathic pulmonary fibrosis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome, granulomatosis with polyangiitis, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis, with the exception of: hypothyroidism (on stable dose of thyroid replacement therapy), asthma managed with inhaled medications only; type 1 diabetes mellitus on stable insulin regimen, Sjögren syndrome, immune thrombocytopenia or autoimmune hemolytic anemia that does not require systemic therapy; dermatologic condition (including eczema, psoriasis, lichen simplex chronicus, or vitiligo) with skin manifestations with rash covering <10% of body surface area and not requiring treatment other than low-potency topical corticosteroids for >12 months prior to registration
13. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
    * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
14. Positive for HIV at screening or any time prior to screening: patients without prior positive HIV test result will undergo an HIV test at screening, unless not permitted under local regulations
15. Active Hepatitis B virus (HBV) infection (chronic or acute): defined as having a positive hepatitis B surface antigen (HBsAg) test at screening. Patients with a past or resolved HBV infection, defined as having a negative HBsAg test and a positive total hepatitis B core antibody test at screening, are eligible for the study
16. Active hepatitis C virus (HCV) infection: defined as positive HCV antibody test followed by a positive HCV RNA test at screening. The HCV RNA test will be performed only for patients who have a positive HCV antibody test
17. Active TB (Mycobacterium tuberculosis)
18. Administration of a live, attenuated vaccine within 28 days before first atezolizumab dose or anticipation that such a live, attenuated vaccine will be required during the study or within 5 months after the final dose of atezolizumab
19. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
20. Inability to swallow medication
21. History of other malignancy that could affect compliance with the protocol or interpretation of results; patients with a curatively treated skin cancer, in situ cervical cancer, or non-CRC malignancy are eligible if the non-CRC malignancy is controlled and will not interfere with measurement of treatment efficacy or safety
22. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 28 days before the first dose of atezolizumab.
23. Any major surgery or significant traumatic injury within 28 days of initiating study treatment or anticipation of need for a major surgical procedure during the study
24. Evidence of other significant or uncontrolled medical or psychiatric conditions that could affect compliance with the protocol
25. Pregnancy, breast-feeding, or prisoner status
26. History of leptomeningeal disease
27. Uncontrolled tumor-related pain
28. Patients requiring pain medication must be on a stable regimen at study entry.
29. Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.

    Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.

    Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).

    • Patients with indwelling catheters (e.g., PleurX) are allowed.
30. Uncontrolled or symptomatic hypercalcemia (ionized calcium 1.5 mmol/L, calcium 12 mg/dL or corrected serum calcium ULN)
31. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.

    • History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
32. Prior allogeneic stem cell or solid organ transplantation
33. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
34. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
To assess the preliminary efficacy with the combination of yttrium-90, capecitabine, and atezolizumab based on the intrahepatic disease control rate (iDCR) at 12 weeks | 12 weeks
  Disease control rate is defined as the proportion of patients with complete response (CR), partial response (PR), or stable disease (SD) within the liver at first post-Y-90 follow-up imaging by NCI's response evaluation criteria in solid tumors (RECIST 1.1), which is a standard way to measure if the tumor is responding to treatment by measuring tumor lesions (cm).

SECONDARY OUTCOMES:
To evaluate the preliminary safety of the combination of yttrium-90, capecitabine, and atezolizumab | Approximately 18 months
  Adverse events will be collected (side effects) per the National Cancer Institute's Common Terminology Criteria for Adverse Events CTCAE v5 (adverse events (side effects) are graded from 1-5).
To determine the extrahepatic disease control rate (eDCR) with the combination of yttrium-90, capecitabine, and atezolizumab | Approximately 18 months
  assessment of extrahepatic disease control rate (eDCR), measurements from up to three of the target lesions identified outside the liver will be utilized to categorize non-liver response according to NCI's response evaluation criteria in solid tumors (RECIST 1.1), which is a standard way to measure if the tumor is responding to treatment by measuring lesions (cm).
To estimate the median overall response rate (ORR), progression free survival (PFS), and overall survival (OS) with the combination of yttrium-90, capecitabine, and atezolizumab | Approximately 18 months
  CT imaging will be performed beginning on Day 90 (+7 days) or Day 132 (+7 days) depending on if the participant received one or two doses of Y-90, respectively. Subsequently, imaging is to be performed every 90 days (+14 days) until disease progression according to NCI's response evaluation criteria in solid tumors (RECIST) 1.1, which is a standard way to measure if the tumor is responding to treatment by measuring lesions (cm).

CONTACTS AND LOCATIONS:
Locations (1):
- Lifespan Cancer Institute: The Miriam and Rhode Island Hospitals Providence, Rhode Island, United States, 02903 Contact:, Providence, Rhode Island, United States